CLINICAL TRIAL: NCT00190723
Title: A Phase II Trial of LY317615 in Patients With Recurrent High-Grade Gliomas
Brief Title: A Study of LY317615 in Patients With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5799; H6Q-MC-JCAJ; NCT00047892 (obsolete NCT alias); NCT00052663 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — enzastaurin

INTERVENTIONS:
Drug: Enzastaurin

SUMMARY:
1. The safety of LY317615 and any side effects that might be associated with the drug.
2. Whether LY317615, can help patients with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* You must be at least 18 years old
* You must have been diagnosed with a recurrent brain tumor by MRI or CT scan
* You must be able to swallow the LY317615 tablets

Exclusion Criteria:

* You are a woman who is pregnant or breastfeeding
* In view of your doctor, you have significant heart, liver, kidney, or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-10; Study Completion 2006-12

PRIMARY OUTCOMES:
To establish data regarding the anti-tumor activity of LY317615 in patients with recurrent high-grade gliomas.

SECONDARY OUTCOMES:
To obtain preliminary information regarding the spectrum of toxicities of LY317615 administered to patients with recurrent high-grade gliomas

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bethesda, Maryland, United States